CLINICAL TRIAL: NCT05020288
Title: A Prospective, Open-label, Multicenter，Single-armed Study of Orelabrutinib in the Treatment of Refractory Primary Immune Thrombocytopenia (ITP)
Brief Title: A Clinical Trial of the Orelabrutinib in the Management of Refractory ITP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITP-Orelabrutinib
Record Dates: First submitted 2021-08-12; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Immune Thrombocytopenia; Bruton's Tyrosine Kinase
Keywords: Orelabrutinib
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — orelabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orelabrutinib (Experimental): Orelabrutinib 50mg po qd
  Interventions: Drug: Orelabrutinib

INTERVENTIONS:
Drug: Orelabrutinib — Orelabrutinib 50mg po qd, every four weeks for one cycle. It will be given three cycles.
  Other Names: ICP-022

SUMMARY:
BTK participates in a variety of signal transduction of innate and adaptive immunity, and has an important role in cell proliferation, differentiation and apoptosis. The impact of BTK inhibitors on hematological malignancies and autoimmune diseases has been well studied. This project was undertaking by Qilu Hospital of Shandong University in China. In order to report the efficacy and safety of the selective BTK inhibitor Orelabrutinib in the management of refractory ITP.

DETAILED DESCRIPTION:
The investigators are undertaking a prospective, open-lable, multicentre trial of 40 refractory ITP adult patients in China. Eligible participants will receive Orelabrutinib in 50 mg po. qd, every 4 weeks for one cycle and it will be given 3 cycles. For non-responders who were well tolerated at 12 weeks of follow-up, the treatment could be extended to 6 cycles. The treatment will be discontinued after 6 months without blood index reaction. In order to report the efficacy and safety of Orelabrutinib in the management of refractory ITP, platelet count, bleeding and other symptoms will be evaluated before and after treatments. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for primary immune thrombocytopenia
* To show a platelet count < 30 * 10^9/L, or with bleeding manifestations, or both
* Willing and able to sign written informed consent
* Meet the diagnostic criteria of refractory ITP according to Chinese guidelines

Exclusion Criteria:

* Secondary thrombocytopenia
* severe immune-deficiency or history of primary immunodeficiency
* active or previous malignancy
* HIV virus infection, tuberculosis, or other active infection (sepsis, pneumonia, or abscess)
* pregnancy or lactation
* diabetes
* hypertension
* cardiovascular diseases
* severe liver or kidney function impairment
* psychosis
* osteoporosis
* inflammatory bowel disease or gastric disease
* arterial or venous thromboembolism within the 6 months before screening or patients who required anticoagulant treatment
* an organ or haematopoietic stem-cell transplantation
* neutrophil count of less than 1500 cells per mm³; glycosylated haemoglobin less than 8%; partial thromboplastin time 1∙5 times or less the upper limit of normal (ULN)
* clinical electrocardiogram changes
* neoplastic disease within the past 5 years
* corrected QT interval greater than 450 ms for men and greater than 470 ms for women;
* substance misuse within the previous 12 months; and those who could not adhere to the protocol or were planning to have a surgical procedure in 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Initial overall response to Orelabrutinib | 14 days after the first dose of Orelabrutinib
  Complete response was defined as a platelet count of 100×10⁹ cells per L or higher and an absence of bleeding. Partial response was defined as a platelet count of 30×10⁹ cells per L or higher, but less than 100×10⁹ cells per L, and at least a doubling of the baseline platelet count and an absence of bleeding. Platelet counts were confirmed on two separate occasions at least 7 days apart when defining complete response or partial response. No response was defined as a platelet count of less than 30×10⁹ cells per L, or less than two-times increase from baseline platelet count, or bleeding.
Sustained overall response to Orelabrutinib | A response lasting for at least 6 months without any additional intervention specific to primary immune thrombocytopenia was defined as a sustained response
  Complete response was defined as a platelet count of 100×10⁹ cells per L or higher and an absence of bleeding. Partial response was defined as a platelet count of 30×10⁹ cells per L or higher, but less than 100×10⁹ cells per L, and at least a doubling of the baseline platelet count and an absence of bleeding. Platelet counts were confirmed on two separate occasions at least 7 days apart when defining complete response or partial response. No response was defined as a platelet count of less than 30×10⁹ cells per L, or less than two-times increase from baseline platelet count, or bleeding.

SECONDARY OUTCOMES:
Time to response | An average of 6 months
  Time from treatment initiation to achieve a complete response or a partial response
Duration of response | through study completion, an average of 1 year
  Time from achievement of a complete response or a partial response to the loss of response (platelet count <30×10⁹ cells per L; measured on two occasions more than 1 day apart or the presence of bleeding).
Therapy associated adverse events | Up to 1 year
  Potential adverse events: leukopenia (report in number * 10^9/L, time of occurrence and duration); nausea and diarrhea (report in frequency); infection (report pathogens and infectious diseases).

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, MD,PhD, Principal Investigator — Shandong University Qilu Hospital